CLINICAL TRIAL: NCT01664533
Title: Prospective, Open-label, Multicenter, National, Non-interventional Phase IV Trial of the Effectiveness, Safety and Tolerability of Tarceva as Second-line Treatment of Patients With Advanced Non-small Cell Lung Cancer (NSCLC), After Failure of First-line Treatment With a Pemetrexed-containing Chemotherapy Regimen
Brief Title: An Observational Study of Erlotinib (Tarceva) as Second-line Treatment in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer After Failure of Pemetrexed in First-line Therapy
Acronym: TIME
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25708
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Erlotinib: Selection of the dose of erlotinib most suitable for each participant was left to the discretion of the physician, guided by the recommendation in the Summary of Product Characteristics. The recommended daily oral dose of erlotinib is 150 mg.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib was supplied as tablets in the retail product Tarceva.
  Other Names: Tarceva

SUMMARY:
This prospective, multicenter observational study will evaluate the efficacy, safety, and tolerability of Tarceva (erlotinib) as second-line treatment in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) who have progressed after pemetrexed-containing first-line chemotherapy. Eligible patients will be followed until withdrawal of consent, lost-to-follow-up, or study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age.
* Histologically or cytologically documented locally advanced or metastatic non-small cell lung cancer (inoperable Stage III or IV according to the 7th TNM Classification of Malignant Tumors).
* Experiencing disease progression after pemetrexed-containing first-line chemotherapy regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Initiated on second-line treatment with Tarceva at the most 4 weeks prior to study entry at baseline (date of signature of informed consent).

Exclusion Criteria:

* Prior chemotherapy/targeted therapy after disease progression after first-line treatment in the advanced non-small cell lung cancer (NSCLC) setting.
* Contraindication for Tarceva according to the Summary of Product characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic non-small cell lung cancer initiated on second-line Tarceva therapy after first-line pemetrexed-containing chemotherapy.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Belgium (21):
  - Aalst
  - Antwerp
  - Boussu
  - Brussels
  - Charleroi
  - Dendermonde
  - Duffel
  - Edegem
  - Frameries
  - Genk
  - Gilly
  - Gosselies
  - Liège
  - Mons
  - Montegnée
  - Namur
  - Ottignies
  - Roeselare
  - Sint-Niklaas
  - Tournai
  - Turnhout

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 59 patients were screened at 17 specialist oncology and pneumology centers in Belgium, 57 of which started Tarceva therapy as second-line treatment and constitute safety analysis (SA) population. Three patients violated the protocol, leaving 54 patients in the per-protocol (PP) population.
Period: Overall Study
Arm/Group | Erlotinib
Started | 57
Completed | 0
Not Completed | 57
Not completed — Death | 42
Not completed — Lost to Follow-up | 3
Not completed — Study termination | 9
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is represented as the per protocol population.
Arm/Group | Erlotinib
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the first dose of erlotinib to disease progression or death from any cause, whichever occurred earlier. Progressive disease was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter of target lesions recorded since treatment started, or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to the end of the study (up to 2 years)
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib
Number analyzed (Participants) | 54
Months | 1.8 [1.4 to 2.6]

2. Secondary Outcome: Best Overall Response
Description: Reported are the percentage of participants with a best overall response of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). The best overall response to treatment was determined by the Response Evaluation Criteria in Solid Tumors (RECIST). A CR was defined as the disappearance of all target lesions (TL) or the disappearance of all non-TLs. A PR was defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD. SD was defined as neither sufficient shrinkage to qualify for a PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD since treatment started for TLs and the persistence of 1 or more non-TL(s). PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since treatment started or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-TLs.
Time Frame: Baseline to the end of the study (up to 2 years)
Population: Per-protocol population: All enrolled participants who started erlotinib therapy and did not violate the study protocol. Only participants with an evaluable response were included in the analysis.
Measure: Number (97.5% Confidence Interval); unit: Percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 52
Percentage of participants
  Complete Response | 0.0 [0.0 to 6.8]
  Partial Response | 0.0 [0.0 to 6.8]
  Stable Disease | 34.6 [21.9 to 49.0]
  Progressive Disease | 65.4 [50.9 to 78.0]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from Baseline until death from any cause.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib
Number analyzed (Participants) | 54
months | 5.8 [3.3 to 8.6]

4. Secondary Outcome: Percentage of Participants Who Developed Rash
Time Frame: Up to 2 years
Population: Safety analysis population: All participants who received at least 1 dose of erlotinib. Data was missing for 1 participant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 56
percentage of participants | 60.7 [46.7 to 73.5]

5. Secondary Outcome: Percentage of Participants Who Developed Diarrhea
Time Frame: Up to 2 years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 56
percentage of participants | 42.8 [29.7 to 56.8]

ADVERSE EVENTS:
Time Frame: Time frame is up to 2 years
Description: Safety analysis population: All participants who received at least 1 dose of erlotinib.
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 17/57
Other Adverse Events (participants affected / at risk) | 51/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=57)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
C-reactive protein increase (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Procalcitonin increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=57)
Rash (Skin and subcutaneous tissue disorders) | 35 (35)
Diarrhea (Gastrointestinal disorders) | 25 (25)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13)
Weight decreased (Investigations) | 8 (8)
Asthenia (General disorders) | 6 (6)
Pyrexia (General disorders) | 5 (5)
Fatigue (General disorders) | 4 (4)
General physical health deterioration (General disorders) | 4 (4)
Chest pain (General disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Conjunctivities (Eye disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.